CLINICAL TRIAL: NCT00613080
Title: A Phase II Evaluation of Preoperative Chemoradiotherapy Utilizing Intensity Modulated Radiation Therapy (IMRT) in Combination With Capecitabine and Oxaliplatin for Patients With Locally Advanced Rectal Cancer
Brief Title: Combination Chemotherapy and Intensity-Modulated Radiation Therapy in Treating Patients Undergoing Surgery for Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0822; CDR0000586277
Record Dates: First submitted 2008-02-09; First posted 2008-02-12 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer
Keywords: stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Radiotherapy; Folfox protocol; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMRT + Chemotherapy , Resection, Postoperative Chemotherapy (Other): Radiation therapy (intensity modulated radiation therapy [IMRT] + three dimensional conformal radiation therapy [3D-CRT]) + neoadjuvant chemotherapy (capecitabine and oxaliplatin) followed by resection and postoperative chemotherapy (FOLFOX)
  Interventions: Drug: capecitabine; Drug: oxaliplatin; Procedure: resection; Radiation: radiation therapy; Drug: FOLFOX

INTERVENTIONS:
Drug: capecitabine — 1650 mg/m^2/day orally 5 days/week during radiotherapy.
Drug: oxaliplatin
  Other Names: 50 mg/m^2 IV over 2 hours weekly for five weeks starting on day 1 of radiotherapy.
Procedure: resection — All patients undergo surgery 4 to 8 weeks following the completion of radiation therapy. The choice of procedure (abdominoperineal resection (APR), low anterior resection (LAR), or LAR/coloanal anastomosis) is at the discretion of the surgeon.
Radiation: radiation therapy — Pelvic intensity modulated radiation therapy (IMRT): 45 Gy in 25 fx Three dimensional conformal radiation therapy (3D-CRT) boost: 5.4 Gy in 3 fx to total dose of 50.4 Gy in 28 fx
Drug: FOLFOX — Postoperative chemotherapy is administered to all patients who have a complete resection of rectal cancer with negative surgical margins and begins within 4-8 weeks following surgical resection, consisting of a total of 9 14-day cycles. Oxaliplatin 85 mg/m^2, IV over 2 hours, day 1.
  Leucovorin 400 mg/m^2, IV over 2 hours, day 1. 5-fluorouracil bolus 400 mg/m^2, IV push, day 1. 5-fluorouracil infusion 2400 mg/m^2, IV continuous infusion over 46 hours, day 1.
  Other Names: Oxaliplatin, leucovorin, 5-fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving these treatments before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects and how well giving combination chemotherapy together with intensity-modulated radiation therapy works in treating patients undergoing surgery for locally advanced rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether the incidence of neoadjuvant acute gastrointestinal toxicity (grade ≥ 2) associated with neoadjuvant chemoradiotherapy is reduced by inverse-planned intensity-modulated radiotherapy (IMRT)-based radiation treatment when compared with conventionally delivered radiotherapy, as was utilized in the capecitabine and oxaliplatin arm of RTOG-0247 (NCT00081289).

Secondary

* To evaluate the feasibility of performing IMRT in a cooperative group setting for the treatment of rectal cancer.
* To estimate the incidence of all toxicity (hematologic and non-hematologic) associated with protocol treatment in the neoadjuvant period, the adjuvant period, and overall.
* To estimate the pathologic complete response rate following neoadjuvant IMRT-based chemoradiotherapy.
* To estimate the time to treatment failure and patterns of failure.
* To correlate pre- and post-treatment levels of serum cytokines with symptoms during and pathological outcomes following neoadjuvant chemoradiotherapy for rectal cancer.
* To evaluate the rate of abdominoperineal resections.

OUTLINE: This is a multicenter study.

* Chemoradiotherapy: Patients undergo inverse-planned intensity-modulated radiotherapy to the pelvis once daily, 5 days a week, for 5 weeks (total of 45 Gy) and a 3-dimensional conformal radiotherapy boost to gross disease once daily for 3 days (total of 45 Gy). Beginning on the first day of radiotherapy and continuing through completion of radiotherapy, patients receive oral capecitabine twice daily, 5 days a week, for 5 weeks and oxaliplatin IV over 2 hours on days 1, 8, 15, 22, 29.
* Surgery: Within 4-8 weeks after completion of chemoradiotherapy, patients undergo resection of the rectal tumor.
* Adjuvant chemotherapy: Beginning 4-8 weeks after surgery, patients with completely resected disease and negative surgical margins receive leucovorin calcium IV over 2 hours and oxaliplatin IV over 2 hours on day 1 and fluorouracil IV bolus on day 1 and fluorouracil IV infusion continuously over 46 hours beginning on day 1 . Treatment repeats every 14 days for up to 9 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months after the start of treatment for 2 years, every 6 months for years 3-5, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed diagnosis of adenocarcinoma of the rectum by biopsy technique that does not completely excise the lesion (e.g., fine needle aspiration, core needle biopsy)

  * Located up to 12 cm from the anal verge with no extension of malignant disease into the anal canal
  * Clinically determined to be stage T3 or T4,N0-N2, and M0 tumor as determined by the following assessments:

    * Colonoscopy and biopsy within 56 days prior to registration
    * History/physical examination (including medication history screen for contraindications) within 56 days prior to registration
    * Contrast-enhanced imaging of the abdomen and pelvis either by computed tomography(CT), MRI, or Positron-emission tomography(PET)-CT (whole body preferred) within 56 days prior to registration
    * Chest x-ray (or CT) of the chest within within 56 days prior to registration to exclude distant metastases (except for patients who have had whole body PET-CT)
    * Transrectal ultrasound (TRUS) within 56 days prior to registration required to establish tumor stage

      * TRUS not required if clinical exam, CT of the pelvis, and/or MRI demonstrates T4 lesion
* No synchronous primary colon carcinoma
* No evidence of distant metastases (M1)

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Zubrod performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,800/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL (transfusion or other intervention to achieve hemoglobin ≥ 8.0 g/dL allowed)
* Aspartate aminotransferase (AST) < 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* Creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior invasive malignancy except nonmelanoma skin cancer unless disease free for a minimum of 3 years

Exclusion criteria:

* Severe, active comorbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 12 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within the past 30 days
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * AIDS
  * Evidence of uncontrolled seizures, central nervous system disorders, or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake
  * Known, existing uncontrolled coagulopathy, unless clinically stable on anticoagulation therapy for ≥ 2 weeks
  * Evidence of peripheral neuropathy ≥ grade 2
* Prior allergic reaction to oxaliplatin or capecitabine
* Lack of physical integrity of the gastrointestinal tract (i.e., severe Crohn disease that results in malabsorption; significant bowel resection that would make one concerned about the absorption of capecitabine) or malabsorption syndrome that would preclude feasibility of oral chemotherapy (i.e., capecitabine)
* Prior systemic chemotherapy for colorectal cancer (prior chemotherapy allowed provided it was for a cancer other than colorectal cancer)
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiotherapy fields
* Major surgery within 28 days of study enrollment(other than diverting colostomy without tumor resection)
* Participation in any investigational drug study within 28 days of study enrollment.
* Concurrent cimetidine, amifostine, and/or depot Sandostatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C. Garofalo, MD, Principal Investigator — University of Maryland Greenebaum Cancer Center; Adam C. Berger, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University; Johanna Bendell, MD, Study Chair — Duke Cancer Institute
Locations (120):
- United States (119):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Auburn Radiation Oncology, Auburn, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Bay Medical, Panama City, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - St. Vincent Oncology Center, Indianapolis, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - St. Peters, City of Saint Peters, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Integris Oncology Services, Oklahoma City, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Upper Delaware Valley Cancer Center, Milford, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- London Regional Cancer Program at London Health Sciences Centre, London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Started | 79
Completed | 68 (Subjects contributing data to the primary analysis are considered to have completed the study.)
Not Completed | 11
Not completed — Ineligible / no protocol treatment | 11

BASELINE CHARACTERISTICS:
Population: All eligible patients.
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Number analyzed (Participants) | 68
Age, Continuous [Median (Full Range); unit: years] | 51 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Experiencing Treatment-related Gastrointestinal Adverse Events ≥ Grade 2 Per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v. 3.0, Occurring Preoperatively
Description: The percentage of patients experiencing preoperative treatment-related gastrointestinal adverse events ≥ grade 2. If patient did not receive surgery, then such adverse events <= 90 days from the start of concurrent treatment are included.
Time Frame: From start of treatment to surgery or ≤ 90 days from the Start of Concurrent Treatment (for patients not undergoing surgery)
Population: Eligible subjects who started study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Number analyzed (Participants) | 68
percentage of patients | 51 [NA to 59] — This is a one-sided confidence interval.
Statistical Analysis 1: Comparison: IMRT + Chemotherapy , Resection, Postoperative Chemotherapy; This study was designed for a one-sided chi-square test to detect at least 12% reduction in the 40% rate of ≥ grade 2 treatment-related preoperative GI AEs from the conventional radiotherapy / capecitabine /oxaliplatin arm of study RTOG-0247 (NCT00081289) with 80% power and a one-sided type I error rate of 0.10; Test type: Superiority or Other; p = 0.93, Chi-squared; Proportion (reported as percentage) = 51

2. Secondary Outcome: Number of Patients in Protocol Adherence Categories for Intensity-modulated Radiotherapy (IMRT) Planning
Description: Real-time quality assurance was performed remotely by the study chair or the radiation oncology co-chair prior to initiation of treatment for the first 40 cases. The final cases enrolled were reviewed within 3 months after accrual was completed. Review included evaluation of clinical target volume (CTV) and planning target volume (PTV), Organs at Risk (OARs), and treatment plan dosimetry.
Time Frame: Pretreatment
Population: Eligible patients who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Number analyzed (Participants) | 68
Participants
  Tumor volume: Contouring score: Per Protocol | 58
  Tumor volume: Contouring score: Acceptable variation | 5
  Tumor volume: Contouring score: Unacceptable variation | 5
  Organs at risk: Contouring score: Per Protocol | 62
  Organs at risk: Contouring score: Acceptable variation | 6
  Organs at risk: Contouring score: Unacceptable variation | 0
  Tumor volume: Dose volume analysis score: Per Protocol | 59
  Tumor volume: Dose volume analysis score: Acceptable variation | 8
  Tumor volume: Dose volume analysis score: Unacceptable variation | 1
  Organs at risk: Dose volume analysis score: Per Protocol | 48
  Organs at risk: Dose volume analysis score: Acceptable variation | 17
  Organs at risk: Dose volume analysis score: Unacceptable variation | 3

3. Secondary Outcome: Number of Patients With Pathologic Complete Response
Description: Pathologic complete response is defined as no evidence of residual cancer histologically in the resection specimen.
Time Frame: At the time of surgery, which is 4-8 weeks after radiation therapy, approximately 9-13 weeks from treatment start.
Population: Eligible patients who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Number analyzed (Participants) | 68
Participants | 10

4. Secondary Outcome: Percentage of Patients With Grade 3 or Higher Treatment-related Adverse Events as Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v3.0
Description: Grade refers to the severity of the adverse event (AE). The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. Adverse events were compiled in four different time periods: 1) Preoperative: Preoperatively or, if no surgery, then ≤ 90 days from the Start of Concurrent Treatment; 2) Postoperative#1: Postoperatively and ≤ 30 days from the Date of Surgery; 3) Postoperative#2: Postoperatively and ≤ 90 days from the End of Postoperative Chemotherapy; 4) Overall: From start of concurrent treatment to end of follow-up;
Time Frame: From study registration to end of follow-up. Maximum follow-up at time of analysis was 5.2 years.
Population: For the four time periods reported, respectively: all registered patients; patients that had surgery; patients that had surgery and postoperative chemotherapy; all registered patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Number analyzed (Participants) | 68
percentage of participants
  Preoperative | 49 [37 to 60]
  Postoperative #1: number analyzed (Participants) | 67
  Postoperative #1 | 7 [3 to 17]
  Postoperative #2: number analyzed (Participants) | 42
  Postoperative #2 | 74 [59 to 85]
  Overall | 78 [67 to 86]

5. Secondary Outcome: Local-regional Failure: 4-year Rate
Description: Local failure is defined as: (1) any recurrence or surgery to the primary site after a complete response (CR) reported at surgery or reported after the end of protocol treatment; or (2) persistence [failure at one day post study entry], absence of CR after protocol treatment was completed and patient lived at least 90 days from the end of treatment. Regional failure is defined as: (1) any recurrence after a nodal CR reported at surgery or reported after the end of protocol treatment; or (2) persistence, absence of nodal CR after protocol treatment was completed and patient lived at least 90 days from the end of treatment. Local-regional failure time is defined as time from registration to local or regional failure, last known follow-up (censored), or death (competing risk). Local-regional failure rates are estimated by the cumulative incidence method.
Time Frame: From registration to four years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Number analyzed (Participants) | 68
percentage of participants | 7.4 [1.0 to 13.7]

6. Secondary Outcome: Distant Failure: 4-year Rate
Description: Distant failure is defined as the appearance of peritoneal seeding or distant metastases. Time to distant failure is defined as time from registration to the date of distant failure, last known follow-up (censored), or death (competing risk). Distant failure rates are estimated by the cumulative incidence method.
Time Frame: From registration to four years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Number analyzed (Participants) | 68
percentage of participants | 29.7 [18.7 to 40.8]

7. Secondary Outcome: Overall Survival: 4-year Rate
Description: Overall survival time is defined as time from registration to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From registration to four years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Number analyzed (Participants) | 68
percentage of participants | 82.9 [70.1 to 90.6]

8. Secondary Outcome: Disease-free Survival: 4-year Rate
Description: Disease is defined as local-regional failure or distant failure. Distant failure is defined as the appearance of peritoneal seeding or distant metastases. Local-regional failure is defined as: (1) any recurrence or surgery to the primary site after a complete response (CR) / any recurrence after a nodal CR - reported at surgery or reported after the end of protocol treatment; or (2) persistence [failure at one day post study entry], absence of primary/nodal CR after protocol treatment was completed and patient lived at least 90 days from the end of treatment. Disease-free survival time is defined as time from registration to the date of disease, death, or last known follow-up (censored). Disease-free survival rates are estimated using the Kaplan-Meier method.
Time Frame: From registration to four years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Number analyzed (Participants) | 68
percentage of participants | 60.6 [47.5 to 71.4]

9. Secondary Outcome: Number of Patients Who Underwent Abdominoperineal Resection
Description: All patients were to undergo surgery 4 to 8 weeks following the completion of radiation therapy. The choice of procedure (abdominoperineal resection (APR), low anterior resection (LAR), or LAR/coloanal anastomosis) was at the discretion of the surgeon. If more than 28 patients received abdominoperineal resection, this would result in a conclusion of an excessive number of abdominoperineal resections.
Time Frame: Surgery occurred 4 to 8 weeks following the completion of radiation therapy, approximately 9-13 weeks from start of treatment.
Population: Eligible patients that had surgery
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Number analyzed (Participants) | 67
Participants | 14

ADVERSE EVENTS:
Description: Eligible patients with adverse event data are included. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy
Serious Adverse Events (participants affected / at risk) | 23/68
Other Adverse Events (participants affected / at risk) | 67/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy (N=68)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Myocardial ischemia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Colonic stenosis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Esophageal hemorrhage (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Rectal hemorrhage (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
Fever (General disorders) | 2
Pain (General disorders) | 1
Peritoneal infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Intraoperative complications (Injury, poisoning and procedural complications) | 1
Rectal anastomotic leak (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Leukopenia (Investigations) | 5
Lymphopenia (Investigations) | 2
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 1
Ischemia cerebrovascular (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash desquamating (Skin and subcutaneous tissue disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT + Chemotherapy , Resection, Postoperative Chemotherapy (N=68)
Blood disorder (Blood and lymphatic system disorders) | 5
Hemoglobin decreased (Blood and lymphatic system disorders) | 40
Vision blurred (Eye disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 25
Anal pain (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 31
Diarrhea (Gastrointestinal disorders) | 55
Dyspepsia (Gastrointestinal disorders) | 9
Dysphagia (Gastrointestinal disorders) | 7
Fecal incontinence (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 11
Mucositis oral (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 48
Proctitis (Gastrointestinal disorders) | 7
Rectal fistula (Gastrointestinal disorders) | 4
Rectal hemorrhage (Gastrointestinal disorders) | 9
Rectal pain (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 25
Chest pain (General disorders) | 8
Chills (General disorders) | 5
Edema limbs (General disorders) | 8
Fatigue (General disorders) | 54
Fever (General disorders) | 10
Pain (General disorders) | 12
Hypersensitivity (Immune system disorders) | 5
Dermatitis radiation (Injury, poisoning and procedural complications) | 13
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 12
Vascular access complication (Injury, poisoning and procedural complications) | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 6
Alanine aminotransferase increased (Investigations) | 24
Alkaline phosphatase increased (Investigations) | 17
Aspartate aminotransferase increased (Investigations) | 23
Creatinine increased (Investigations) | 6
Hyperbilirubinemia (Investigations) | 11
Laboratory test abnormal (Investigations) | 6
Leukopenia (Investigations) | 41
Lymphopenia (Investigations) | 23
Neutrophil count decreased (Investigations) | 34
Platelet count decreased (Investigations) | 34
Weight loss (Investigations) | 18
Anorexia (Metabolism and nutrition disorders) | 27
Dehydration (Metabolism and nutrition disorders) | 18
Hyperglycemia (Metabolism and nutrition disorders) | 35
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 16
Hypocalcemia (Metabolism and nutrition disorders) | 20
Hypokalemia (Metabolism and nutrition disorders) | 17
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Joint pain (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 13
Neurological disorder NOS (Nervous system disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 8
Peripheral sensory neuropathy (Nervous system disorders) | 50
Taste alteration (Nervous system disorders) | 15
Agitation (Psychiatric disorders) | 5
Anxiety (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 22
Cystitis (Renal and urinary disorders) | 6
Urinary frequency (Renal and urinary disorders) | 13
Urinary incontinence (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 8
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 12
Rash desquamating (Skin and subcutaneous tissue disorders) | 10
Skin disorder (Skin and subcutaneous tissue disorders) | 5
Sweating (Skin and subcutaneous tissue disorders) | 6
Hot flashes (Vascular disorders) | 6
Hypotension (Vascular disorders) | 5
Thrombosis (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No